CLINICAL TRIAL: NCT00366457
Title: Phase II Study of Gemcitabine, Bevacizumab and Erlotinib in Locally Advanced and Metastatic Pancreatic Cancer
Brief Title: Gemcitabine, Bevacizumab and Erlotinib in Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry); Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Lawrence S. Blaszkowsky, MD, Assistant Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-234
Record Dates: First submitted 2006-08-17; First posted 2006-08-21 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-04

CONDITIONS: Pancreatic Cancer; Adenocarcinoma of the Pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Bevacizumab and Erlotinib (Other): single-arm, no masking
  Interventions: Drug: Bevacizumab; Drug: Erlotinib; Drug: Gemcitabine

INTERVENTIONS:
Drug: Bevacizumab — Given intravenously on days 1 and 25 of every 28-day cycle (one every 2 weeks). Participants may continue to receive study treatment as long as there is no disease progression or serious side effects.
  Other Names: rhuMAb VEGF
Drug: Erlotinib — Taken orally every day. Participants may continue to receive study treatment as long as there is no disease progression or serious side effects.
  Other Names: Tarceva
Drug: Gemcitabine — Given intravenously on days 1, 8 and 15 of each 28-day cycle. Participants may continue to receive study treatment as long as there is no disease progression or serious side effects.
  Other Names: Gemzar

SUMMARY:
The main purpose of this study is to learn whether or not the combination of gemcitabine, bevacizumab and erlotinib works in treating patients with advanced or metastatic pancreatic cancer. Bevacizumab is a new anti-cancer drug. It is an antibody that works to slow or stop cell growth in cancerous tumors by decreasing the blood supply to the tumors. It is approved by the FDA for the treatment of colorectal cancer but is still considered investigational for treating pancreatic cancer.

DETAILED DESCRIPTION:
* Participants will receive study treatment as an outpatient. The study treatment will be given in time periods called cycles. Each treatment cycle will be 28 days.
* Gemcitabine will be given intravenously on days 1, 8, and 15 (once per week for the first three weeks) of the treatment cycle.
* Bevacizumab will be given intravenously on days 1 and 15 (once every 2 weeks) of the treatment cycle.
* Erlotinib will be taken orally every day of the treatment cycle.
* Participants will see the doctor or nurse practitioner every week for the first 28 days of treatment. During all of the following cycles, they will see the doctor or nurse practitioner on day 1 and day 15 of each cycle.
* Each 4-week cycle can be repeated until the participant or the doctor decided that they should be removed from the study.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with unresectable or metastatic adenocarcinoma of the pancreas
* ECOG Performance Status 0-2
* 18 years of age or older
* Radiographically measurable disease
* Expected survival of at least 4 months
* Creatinine of </= 2.0
* Adequate hepatic function
* Adequate hematopoietic function
* Use of effective means of contraception in subjects of child-bearing potential

Exclusion Criteria:

* Warfarin anticoagulation
* Prior treatment with a tyrosine kinase inhibitor, EGFR inhibitor, or VEGF inhibitor
* Coexistent malignant disease
* Current or recent (within 4 weeks) participation in a clinical trial
* Pregnancy
* Documented invasion of adjacent organs or major blood vessels
* Blood pressure of > 150/100mmHg
* Unstable angina
* NYHA Grade II or greater congestive heart failure
* History of myocardial infarction or stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis of coagulopathy
* Presence of CNS or brain metastases
* Major surgical procedure, open biopsy, or significant traumatic event within 28 days
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months
* Serious non-healing wound, ulcer or bone fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08; Primary Completion 2008-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence S. Blaszkowsky, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Started | 32
Completed | 30
Not Completed | 2
Not completed — never began study therapy | 2

BASELINE CHARACTERISTICS:
Population: participants who started treatment
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression
Description: Time to tumor progression (TTP) = time from date of initial treatment to first objective documentation of progressive disease or death; patients who die without a reported prior progression will be considered to have progressed on the day of their death.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: all patients will be followed for a minimum of 4 months
Population: participants who started treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Number analyzed (Participants) | 30
months | 3.5 [2.6 to 5.6]

2. Secondary Outcome: Response Rate
Description: Response rate using RECIST criteria and latest time point available. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: after at least one 28-day cycle of treatment
Population: participants with response data available
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Number analyzed (Participants) | 28
Participants
  Partial Response | 1
  Progressive Disease | 8
  Stable Disease | 19

3. Secondary Outcome: Toxicity Profile
Description: Grade 3-4 treatment-related toxicities (treatment-related = possible, probable, or definite) Grading system: 1= mild, 2 = moderate, 3 = severe, 4 = life-threatening
Time Frame: during and after first 28-day cycle of treatment
Population: participants who started treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Number analyzed (Participants) | 30
Participants
  Neutrophils | 4
  ALT-SGPT | 3
  Fatigue | 2
  Leukocytes | 2
  Rash: acne/acneiform | 2
  Thrombosis/thrombus/embolism | 2
  Anorexia | 1
  AST - SGOT | 1
  Hemoglobin | 1
  Lymphopenia | 1
  Nonneuropathic generalized weakness | 1
  Upper GI-hemorrhage NOS | 1
  Vascular access-Thrombosis/embolism | 1
  Vessel injury - artery - Other NOS | 1
  Weight loss | 1

4. Secondary Outcome: Overall Survival
Description: overall survival (OS) = time from study entry until death from any cause
Time Frame: 5 years
Population: participants who started treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Number analyzed (Participants) | 30
months | 6.7 [4.9 to 11.7]

ADVERSE EVENTS:
Arm/Group | Gemcitabine, Bevacizumab and Erlotinib
Serious Adverse Events (participants affected / at risk) | 11/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Bevacizumab and Erlotinib (N=30)
Pumonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Death from disease progression (Endocrine disorders) | 3 (3)
Death from infection or sepsis (Infections and infestations) | 2 (2)
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1 (1)
Brain Infarct (Nervous system disorders) | 1 (1)
Neutropenia (Immune system disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Bevacizumab and Erlotinib (N=30)
Fatigue (General disorders) | 25 (102)
Leukocytes (Blood and lymphatic system disorders) | 25 (84)
Nausea (Gastrointestinal disorders) | 24 (73)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 23 (91)
Hyperglycemia (Metabolism and nutrition disorders) | 23 (71)
Platelets (Blood and lymphatic system disorders) | 22 (80)
ALT- SGPT (Metabolism and nutrition disorders) | 22 (76)
Hemoglobin (Blood and lymphatic system disorders) | 21 (78)
Neutrophils (Blood and lymphatic system disorders) | 21 (67)
AST- SGOT (Metabolism and nutrition disorders) | 20 (77)
Abdomen - pain (General disorders) | 20 (47)
Anorexia (Gastrointestinal disorders) | 19 (48)
Constipation (Gastrointestinal disorders) | 17 (34)
Hyponatremia (Metabolism and nutrition disorders) | 17 (27)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 16 (61)
Weight loss (General disorders) | 15 (35)
Vomiting (Gastrointestinal disorders) | 15 (25)
Rigors/chills (General disorders) | 15 (20)
Lymphopenia (Blood and lymphatic system disorders) | 14 (30)
Alkaline phosphatase (Metabolism and nutrition disorders) | 13 (25)
Nose- hemorrhage (General disorders) | 11 (19)
Fever w/o neutropenia (General disorders) | 11 (12)
Bilirubin (Metabolism and nutrition disorders) | 10 (19)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (24)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (15)
Insomnia (General disorders) | 9 (14)
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 8 (9)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 7 (13)
Skin-other (Skin and subcutaneous tissue disorders) | 7 (12)
Dehydration (Gastrointestinal disorders) | 7 (9)
Head/headache (General disorders) | 6 (13)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 (12)
Muco/stomatitis by exam- oral cavity (Gastrointestinal disorders) | 6 (10)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (8)
Extremity-limb- pain (General disorders) | 6 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (23)
Hypertension (Cardiac disorders) | 5 (22)
Proteinuria (Metabolism and nutrition disorders) | 5 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (13)
Depression (Nervous system disorders) | 5 (11)
Flatulence (Gastrointestinal disorders) | 5 (10)
Edema limb (Blood and lymphatic system disorders) | 5 (9)
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Bicarbonate (Metabolism and nutrition disorders) | 5 (6)
Hypokalemia (Metabolism and nutrition disorders) | 5 (5)
Muscle- pain (General disorders) | 5 (5)
GI-other (Gastrointestinal disorders) | 4 (7)
Back- pain (General disorders) | 4 (6)
Dizziness (Nervous system disorders) | 4 (6)
Infection Gr0-2 neut- upper airway (Infections and infestations) | 4 (5)
Chest/thoracic pain NOS (General disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (10)
Neurologic-other (Nervous system disorders) | 3 (6)
Allergic reaction (Immune system disorders) | 3 (4)
Anxiety (Nervous system disorders) | 3 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4)
Pain-other (General disorders) | 3 (4)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Throat/pharynx/larynx- pain (General disorders) | 3 (4)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Ocular-other (Eye disorders) | 3 (3)
Pain NOS (General disorders) | 3 (3)
Taste disturbance (Gastrointestinal disorders) | 3 (3)
Distention/bloating- abdominal (Gastrointestinal disorders) | 2 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (4)
Neuropathy-sensory (Nervous system disorders) | 2 (3)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2)
Burn (Skin and subcutaneous tissue disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (2)
Flu-like syndrome (General disorders) | 2 (2)
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2)
Joint- pain (General disorders) | 2 (2)
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 2 (2)
Rectum- hemorrhage (General disorders) | 2 (2)
Rectum- pain (General disorders) | 2 (2)
Renal/GU-other (Renal and urinary disorders) | 2 (2)
Sweating (General disorders) | 2 (2)
Thrombosis/thrombus/embolism (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes